CLINICAL TRIAL: NCT03361488
Title: Effect of Structured Patient Interviews in the Preoperative Anesthesia Clinic on Recall of Relevant Information
Acronym: SPI-RECALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolai Goettel (Other)
Responsible Party: Sponsor-Investigator, Nicolai Goettel, MD, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SPI-RECALL
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Anesthesia; Surgical Procedure, Unspecified; Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trained anesthesiologist (Experimental): Patient interview by anesthesiologists having obtained training to optimize structured communication
  Interventions: Other: Trained anesthesiogist
- Control anesthesiologist (No Intervention): Patient interview by control anesthesiologists

INTERVENTIONS:
Other: Trained anesthesiogist
  Arms: Trained anesthesiologist

SUMMARY:
The preanesthetic visit influences patient satisfaction and medical outcome. This study aims to evaluate whether training for a structured interview technique improves communication skills, resulting in increased recall of relevant information by surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients in the preoperative anesthesia clinic
* Written informed consent

Exclusion Criteria:

* Inadequate comprehension of the German language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Recall of information | Immediately after patient interview
  Number of recalled information items in free text, expert assessment according to predefined Delphi criteria

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Goettel, MD, Principal Investigator — University Hospital, Basel, Switzerland; Albert Urwyler, MD, Study Chair — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland